CLINICAL TRIAL: NCT04609293
Title: Observational Study of Camrelizumab Combined With Apatinib and Hyperfractionated Radiotherapy for Renal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Xian-shu Gao, Professor, Peking University First Hospital
Other Study IDs: 20200903
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Camrelizumab+apatinib+Hypofractionated radiation therapy: Camrelizumab:200mg every 2 weeks for 1 years or until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
  Apatinib:250mg everyday until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment.
  Radiation: one week following completion of the second immunotherapy, hypofractionated radiotherapy with marginal dose of 50Gy/2Gy/25f and tumor center dose of local hyperfraction increase 24-32Gy/8-12Gy/3-4f will be performed 3-5 times. The routine radiotherapy will be started at the same time as the third immunotherapy and 25 times routine radiotherapy will be completed before the fifth or sixth immunotherapy.
  Interventions: Combination Product: camrelizumab+apatinib+hyperfractionated radiotherapy

INTERVENTIONS:
Combination Product: camrelizumab+apatinib+hyperfractionated radiotherapy — Immunotherapy, anti-angiogenesis targeted therapy combined with hyperfractionated radiotherapy

SUMMARY:
This trial will explore effectiveness and safety using the combination therapy of camrelizumab，apatinib and hyperfractionated radiotherapy in patients with renal cell carcinoma(RCC). Hypofractionation is a technique that delivers higher daily doses of radiation over a shorter period of time.immunotherapy. hyperfractionated radiotherapy, represented by stereotactic body radiation therapy (SBRT), can significantly improve the radiotherapy sensitivity of RCC. This trial will also observe whether SBRT can bring about immune effects and explore the group and individual indicators that affect the treatment effect of RCC.

DETAILED DESCRIPTION:
This trial is a prospective, single-center, observational clinical trial evaluating the combination therapy of camrelizumab，apatinib and hyperfractionated radiotherapy in patients with renal cell carcinoma(RCC). All enrolled patients will receive the following treatments: camrelizumab 200mg every 2 weeks for 1 years combined with apatinib 250mg everyday until disease progression (as determined by RECIST 1.1), intolerance, or patient/physician decision to stop treatment. One week following completion of the second immunotherapy, hypofractionated radiotherapy with marginal dose of 50Gy/2Gy/25f and tumor center dose of local hyperfraction increase 24-32Gy/8-12Gy/3-4f will be performed 3-5 times. The routine radiotherapy will be started at the same time as the third immunotherapy and 25 times routine radiotherapy will be completed before the fifth or sixth immunotherapy.

During treatment participants will be assessed for curative effects and the occurrence of adverse events. Following treatment, participants will be assessed at a clinic visit every 3 months to collect survival information and follow-up treatment information. The planned sample size is 30 study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with clear cell renal cell carcinoma were confirmed by histological or cytological;
2. Locally advanced/metastatic (the newly diagnosed stage IV RCC assessed by AJCC) or recurrent RCC;
3. Have not received or received systemic treatment for first-line advanced HCC (including but not limited to a variety of targeted therapies including TKI, VEGF and mTOR);
4. The number of measurable lesion is not more than 5, or although the number of measurable lesion is more than 5, but the radiotherapy department and imaging doctors evaluate that the measurable lesions that can accept radiotherapy are more than or equal to 3;
5. According to RECIST 1.1 standard, there will be clinically assessable lesions, and the target lesion has not received radiotherapy before;
6. Male or female,from 18 to 75 years;
7. The life expectancy will be longer than 6 months;
8. ECOG score will be 0 - 2;
9. The main organ functions are normal, and there is no serious blood, heart, lung, liver, kidney dysfunction and immune deficiency diseases. The results of laboratory test must be met the following criteria: Neutrophils: more than 1.5 × 109/L; ; Platelets: more than 100 × 109/L; Hemoglobin: more than 100g/L; serum albumin：more than 30 g/L; bilirubin：less than the upper normal limit (ULN); ALT and AST：less than 2.5 folds of the upper normal limit (ULN)，if there is liver metastasis, ALT and AST must be less than 5 folds of the upper normal limit (ULN) ; Serum Creatinine: less than 1.5×ULN; Blood Urea Nitrogen (BUN): less than 2.5×ULN; Thyroid Stimulating Hormone (TSH): ess than the upper normal limit (ULN)，if abnormal, the T3 and T4 levels should be examined, and the T3 and T4 levels are normal;
10. Be willing to comply with research and follow-up procedures;
11. Female and male subjects should take effective contraceptive measures from the beginning of treatment to within 6 months after the end of treatment.Agreeing to participate in this study and signing a written informed consent.

Exclusion Criteria:

1. Central nervous system metastasis (including brain metastasis, meningeal metastasis, etc.);
2. Other immunosuppressive drugs used within 14 days before before study drug administration, excluding nasal sprays and inhaled corticosteroids or physiological doses of systemic steroids (ie not more than 10 mg/day of prednisolone or Other corticosteroids of equivalent pharmacological physiological dose);
3. Hypertension and unable to be controlled within normal level following treatment of anti-hypertension agents: systolic blood pressure ≥140 mmHg, diastolic blood pressure ≥ 90 mmHg;
4. Clinically significant cardiovascular diseases：Myocardial ischemia or myocardial infarction above grade II, ventricular arrhythmia which poorly controlled，QTc>450ms（male）/QTc>470ms (female)；Congestive heart failure (New York heart association (NYHA) class is Ⅲ～Ⅳ)；or cardiac color Doppler ultrasound examination revealed that the left ventricular ejection fraction (LVEF) <50%;
5. Accompanied by uncontrolled pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
6. Patients with any active autoimmune disease or history of autoimmune disease, including but not limited to the following: hepatitis, pneumonitis, uveitis, colitis (inflammatory bowel disease), hypophysitis, vasculitis, nephritis, hyperthyroidism, and hypothyroidism;
7. Asthma that requires intermittent use of bronchodilators or other medical intervention should be excluded（Asthma has been completely relieved in childhood, and those without any intervention after adulthood can be included）;
8. Coagulation abnormalities (INR>1.5、PT>ULN+4s、APTT >1.5 ULN）, with bleeding tendency or are receiving thrombolytic or anticoagulant therapy;
9. Proteinuria ≥ (++) and 24 hours total urine protein > 1.0 g;
10. Received major surgery or suffered severe traumatic injury, fracture or ulcer within 4 weeks before enrollment;
11. Severe infections (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) within 4 weeks before the first administration, or unexplained fever> 38.5°C during the screening period/before the first administration;
12. Clinically significant hemoptysis or more than half a teaspoon (2.5ml) of hemoptysis per day occurred within 2 months before enrollment; or Clinically significant bleeding symptoms or tendency, such as gastrointestinal bleeding, hemorrhagic Gastric ulcer, fecal occult blood≥++ at baseline, or vasculitis, etc.;
13. Arterial/venous thrombosis events occurred in the 12 months before enrollment, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
14. History of immunodeficiency or human immunodeficiency virus (HIV) infection: HBV DNA>500 IU/ml, HCV RNA>1000copies/ml, HBsAg+ and anti-HCV+；
15. Has a known additional malignancy within the last 5 years, exceptions include basal cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer;
16. The patient is using other research or standard anti-tumor drugs;
17. Patients with a clear history of allergies may be potentially allergic or intolerant to camrelizumab and apatinib;
18. Patients who have a history of psychotropic drug abuse and cannot be quit or have mental disorders;
19. Other condition, illness, psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or stereotactic radiotherapy administration, or may interfere with the interpretation of study results and in the judgment of the investigator would make the patient inappropriate for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous sampling was performed in the Department of Radiotherapy, Peking University First Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-10-20 (Estimated); Primary Completion 2023-09-07 (Estimated); Study Completion 2024-05-07 (Estimated)

PRIMARY OUTCOMES:
Objective response rate（ORR） | 3 years
  Objective response rate, which is defined as the proportion of subjects who achieve a best response of complete response (CR) or partial response (PR) using the RECIST 1.1 criteria.

SECONDARY OUTCOMES:
Subject safety | Date of signing of informed consent form until 12 weeks after the last medication
  Number of Adverse Events using NCI CTCAE 5.0
Progression free survival (PFS) | 3 years
  The date of first treatment until the date of progression using the RECIST 1.1 criteria, or death due to any cause, whichever comes first.
Disease control rate(DCR) | 3 years
  Disease control rate, which is defined as the proportion of subjects who achieve a response of complete response，partial response and stable disease (PR+CR+SD) in the total number of evaluable subjects using the RECIST 1.1 criteria.
Overall Survival(OS) | 3 years
  Overall survival, defined from the date of first treatment to the date of death due to any cause.
Local Control Rate | 3 years
  Local Control Rate, which is defined as the proportion of subjects who achieve a response of remission and stable disease (PR+CR+SD) evaluated by RECIST 1.1 after radiotherapy.
Quality of Life: EORTC QLQ-C30 questionnaire | 3 years
  Quality of life, which will be evaluated using the EORTC（The European Organization for Reasearch and Treatment of Cancer） QLQ-C30（Quality of Life Questionnare-Core 30） questionnaire. The questionnaire contains 30 items. Items 29 and 30 are divided into seven levels, which are counted from 1 to 7 points, 1 is very poor, and 7 is very good. Other items are divided into 4 levels: no at all, a little bit, a lot, and very, and they are directly rated from 1 to 4 points.
Response rate of lesions that did not receive radiotherapy | 3 years
  Response rate of lesions that did not receive radiotherapy, which is defined as the percentage of the number of cases with tumors that have not received radiotherapy in remission and stable disease (PR+CR+SD) in the total number of evaluable cases using the RECIST 1.1 criteria.
Pathology and genetic testing | 3 years
  The pathology of the primary tumor before treatment, the puncture specimen of the tumor after the end of radiotherapy, and the whole exome sequencing of the tumor pathology after the progression + blood ctDNA detection for the patients who agree to the examination.

CONTACTS AND LOCATIONS:
Overall Officials: Xianshu Gao, MD,PhD, Principal Investigator — Peking University First Hospital

IPD SHARING:
Plan to Share IPD: No